CLINICAL TRIAL: NCT04023344
Title: An Open-label, Randomized, Multi-center, Parallel-group Clinical Trial Comparing the Efficacy and Safety of Insulin Lispro Biphasic 25 ("Geropharm", Russia) Humalog® Mix 25 ("Lilly France", France) in Type 2 Diabetes Mellitus Patients
Brief Title: Efficacy and Safety of Insulin Lispro Biphasic 25 Compared to Humalog® Mix 25 in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LISPRO25-IM
Record Dates: First submitted 2019-07-05; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-01

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 2; Lispro Biphasic; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — insulin lispro, isophane insulin lispro drug combination (25:75)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Humalog® Mix 25 (Active Comparator): Insulin Humalog® Mix 25 twice daily, individually glucose-level based administered doses +/- 1 or 2 OADs in stable doses, started before enrollement
  Interventions: Drug: Humalog Mix25
- Insulin Lispro Biphasic 25 (Experimental): Insulin Lispro Biphasic 25 twice daily, individually glucose-level based administered doses +/- 1 or 2 OADs in stable doses, started before enrollement
  Interventions: Drug: Insulin Lispro Biphasic 25

INTERVENTIONS:
Drug: Humalog Mix25 — Subcutaneus injections Humalog® Mix 25 twice daily during 4 weeks of glucose-level based dose titration, 24 weeks of treatment with stable doses
  Arms: Humalog® Mix 25
Drug: Insulin Lispro Biphasic 25 — Subcutaneus injections Insulin Lispro Biphasic 25 ("Geropharm") twice daily during 4 weeks of glucose-level based dose titration, 24 weeks of treatment with stable doses
  Arms: Insulin Lispro Biphasic 25

SUMMARY:
The study is designed to approve non-inferior efficacy and safety of Insulin Lispro Biphasic 25 ("Geropharm") compared to Humalog® Mix 25 in Type 2 Diabetes Mellitus Patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed written consent
* Clinical diagnosis of type 2 diabetes mellitus for at least 6 months prior to screening
* Glycosylated hemoglobin (HbA1c) level of 7.6 to 12.0 % at screening (both values inclusive)
* Body mass index (BMI) of 18.0 to 35 kg/m2 at screening (both values inclusive)
* Stable doses OADs for at least 3 months prior to treatment of experimental drug
* Female patients of childbearing potential who are willing to use two acceptable methods of contraception, (e.g., intra-uterine device plus condom, spermicidal gel plus condom, diaphragm plus condom, etc.), from the time of screening and for the duration of the trial, through trial completion

Exclusion Criteria:

* Acute inflammation disease for 3 weeks prior to screening
* Deviation of the laboratory results conducted during the screening:

Hemoglobin value < 9,0 g/dl; Hematocrit value < 30 %; ALT and AST value > 2 folds as high as maximal normal value; Serum bilirubin value > 1.5 folds as high as maximal normal value

* History of hematological disorders that can affect the reliability of HbA1c estimation (hemoglobinopathies, hemolytic anemia, etc.)
* Serious blood loss for 3 months prior to screening (blood donation, surgery procedure, etc.)
* Contraindication to the use of insulin Lispro Biphasic 25
* Insulin resistance over 1.5 U/kg insulin pro day
* Presence of insulin antibodies in the blood at the screening ˃10 U/ml
* Use of 3 or more oral antidiabetic drugs (OAD)
* Presence of severe diabetes complications
* History or presence of uncontrolled diabetes mellitus for 6 months prior to screening
* Deviation of vital signs, which can influence to results
* History of administration of glucocorticoids for 1 year prior to screening
* History of autoimmune disease, except controlled autoimmune thyroid disease
* Pregnant and breast-feeding women
* History of hypersensitivity to any of the active or inactive ingredients of the insulin/insulin analogue preparations used in the trial, OR history of significant allergic drug reactions
* Administration of any immunosuppressive drugs (Cyclosporinum, Methotrexatum)
* Incomplete recovery after surgery procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
Antibody Response | 26 weeks
  Change from baseline in titer of antibodies to human insulin

SECONDARY OUTCOMES:
Adverse Events frequency and degree | 26 weeks (4+22 weeks)
  Hypoglycemic episodes (glucose level < 3.9 mmol/l) frequency Occurrence of local reactions at injection sites Occurrence allergic reactions
HbA1c | 26 weeks
  Change in HbA1c from baseline
Fasting Plasma Glucose Level | 26 weeks
  Change in fasting plasma glucose level from baseline
Seven-Point Glucose Testing | 26 weeks
  Change in seven-point glucose testing results from baseline
Insulin Dose | 26 weeks
  Change in total insulin dose per body weight (U/kg) from baseline
Body Mass Index | 26 weeks
  Change in BMI from baseline
Treatment Satisfaction | 26 weeks
  Change in overall treatment satisfaction (DTSQ score) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandr Yu Mayorov, MD, Principal Investigator — Endocrinology Research Centre
Locations (18):
- Russia (18):
  - Chelyabinsk Railway Clinical Hospital, Chelyabinsk
  - Railway Clinical Hospital N.A. Semashko, Moscow
  - Endocrinology Research Centre (Moscow), Moscow
  - Moscow Endocrinological Dispensary, Moscow
  - Nizhny Novgorod Regional Clinical Hospital, Nizhny Novgorod
  - V.A. Baranov Republic Hospital, Petrozavodsk
  - Rostov State Medical University, Rostov-on-Don
  - City Polyclinic № 77, Saint Petersburg
  - City Hospital № 2, Saint Petersburg
  - City Polyclinic № 117, Saint Petersburg
  - City Polyclinic № 17, Saint Petersburg
  - Institute of Medical Research, Saint Petersburg
  - Research Center Eco-Safety, Saint Petersburg
  - City Hospital №40, Saint Petersburg
  - Pokrovskaya Municipal Hospital, Saint Petersburg
  - Diabetes Center, Samara
  - Clinical City Hospital № 9, Saratov
  - Siberian State Medical University, Tomsk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayorov AY, Mosikian AA, Alpenidze DN, Makarenko IE, Orlova VL, Lunev IS, Verbovaya MV, Zinnatulina BR, Khokhlov AL, Drai RV. Efficacy and safety of GP40021 insulin lispro biphasic compared with Humalog Mix 25 in Type 2 diabetes mellitus patients. J Comp Eff Res. 2021 Jan;10(1):55-66. doi: 10.2217/cer-2020-0064. Epub 2020 Dec 23. PMID 33355484